CLINICAL TRIAL: NCT06802289
Title: Preventing Frailty in Hospital Through Mobilizing Patients: a Pilot RCT
Brief Title: Preventing Frailty in Hospital Through Mobilizing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Vitalite Health Network (Unknown)
Responsible Party: Principal Investigator, Myles William O'Brien, Dr., Université de Sherbrooke
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 102088
Record Dates: First submitted 2024-11-21; First posted 2025-01-31 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Frailty At Older Adults
Keywords: Frailty management; Mobilization; Sex differences; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Males (Experimental): A team of Kinesiologists visit the patients daily from admission to discharge to promote movement and help them mobilize to the best of their capabilities (e.g., walking, standing, or sitting on the edge of the bed).
  Interventions: Behavioral: Mobility promotion
- Females (Experimental): A team of Kinesiologists visit the patients daily from admission to discharge to promote movement and help them mobilize to the best of their capabilities (e.g., walking, standing, or sitting on the edge of the bed).
  Interventions: Behavioral: Mobility promotion

INTERVENTIONS:
Behavioral: Mobility promotion — At the Georges-L. Dumont hospital, a patient mobilization program has been introduced on floor 4C that embeds Kinesiologists within care to visit patients daily. A team of Kinesiologists visit the patients daily to promote movement and help them mobilize to the best of their capabilities (e.g., walking, standing, or sitting on the edge of the bed). The investigators propose to continue this individualized model but incorporate activity and frailty measures in males and females older adults.

SUMMARY:
Frailty describes the variability in aging and explains why two people of the same chronological age may look very different. Higher frailty leads to poor quality of life, disability, and death. Hospitalized patients living with frailty have a higher risk for functional decline, new impairments in activities of daily living, a longer hospital stay, hospital readmission, and death. A previous study from our team has reported that 60% of inpatients have more difficulty with 1+ basic activity of daily living (i.e., eating, getting out of bed, using the toilet, etc.) after hospitalization compared to pre-admission, with 1-in-4 patients having difficulty with 3+ basic tasks. Patients with few health deficits can recover to their pre-admission level, but those with higher frailty levels cannot, priming them for readmissions. Physical activity and reducing time spent sitting or lying postures prevent and improve frailty. Older patients who walk at least once/day outside their room during hospitalization have ~1.7 days shorter length of hospital stay compared with those who stayed in their room. Although multiple barriers exist to promoting upright time in a hospital, strategies that help address patients' excessive time spent in bed are often not implemented but could attenuate the development of frailty in the hospital. Few exercise interventions in hospital studies have considered frailty. The investigators have conducted a clinical trial within the Halifax Infirmary (Nova Scotia Health) that focused on mobilizing patients (average age: ~75 years) via regular visits by a Kinesiologist and observed that the intervention groups reduced their frailty level from preadmission and admission versus discharge. While preliminary findings from this model were promising, its reach was limited to acute geriatric care and dependent upon researchers to conduct the intervention. At the Georges-L. Dumont hospital, a patient mobilization program has been introduced in General and Internal Medicine (floor 4C) that embedded Kinesiologists within care to visit patients daily. Preliminary findings indicate that patients and staff are enjoying the program via self-report questionnaire. However, evaluations of the program's effectiveness in changing objectively measured activity and frailty levels and whether multiple patient visits would be more effective (e.g., refining the program) are unclear. The investigators propose to evaluate the effectiveness of the existing patient mobilization program and if more patient contact improves outcomes. Our study integrates activity monitoring technology and frailty assessments to help patients leave the hospital healthier and decrease the risk of readmission. Study Objectives: The proposed study will test the hypothesis that, compared to usual care (Kinesiology visit once/day), patients who receive multiple check-ins will, 1) increase their step counts and upright time, 2) decrease their frailty level, and 3) have a less length of stay and less readmission rates.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients are:

1. 50 years or older,
2. projected to be in-hospital for at least 3-days,
3. not in a shared room with another study participant, and
4. can independently provide consent or have a caregiver to provide consent.

Exclusion Criteria:

* Patients enrolled in other clinical trials or interventions that might confound the results of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Severity of Frailty | At enrollment and at the end of treatment, approximately 2 weeks
  Frailty will be assessed in each participant using the validated Frailty Index used extensively by our group, which calculates frailty as a proportion of health problems present in each person. A trained researcher will help the patient complete the Frailty Index and measure participants' frailty using the Clinical Frailty Scale (scored from 1 [very fit] to 9 [terminally ill]). This scale ensures us a way to obtain a graded frailty score for participants who might be unable to complete the longer questionnaire with assistance.
Accumulation of Physical Activity & Postures in Hospital | From enrollment through to the end of treatment, approximately 2 weeks
  Movement will be measured using activPAL inclinometers positioned on the patients' torso, thigh, and shin. Monitors will be waterproofed and attached 24-hr/day for at least 3-days using a clear medical dressing. We have safely attached these devices to patients' skin for longer durations (14+ days). Physical activity (step counts, physical activity intensity), upright posture, and detailed sedentary postures (e.g., sitting versus lying time) will be determined via validated, custom software that was developed and openly published by our group.

SECONDARY OUTCOMES:
Hospital Length of Stay | This will be derived at discharge of patient from the hospital (at least 3-days)
Rate of Hospital Readmissions | Hospital readmissions within 30 days will be quantified by medical records one-month after hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Georges-L.-Dumont University Hospital Centre, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to concerns related to participant confidentiality and privacy. As a result, we have decided not to make the data publicly available.

REFERENCES:
- [Background] Afilalo J, Karunananthan S, Eisenberg MJ, Alexander KP, Bergman H. Role of frailty in patients with cardiovascular disease. Am J Cardiol. 2009 Jun 1;103(11):1616-21. doi: 10.1016/j.amjcard.2009.01.375. Epub 2009 Apr 8. PMID 19463525
- [Background] Theou O, Kehler DS, Godin J, Mallery K, MacLean MA, Rockwood K. Upright time during hospitalization for older inpatients: A prospective cohort study. Exp Gerontol. 2019 Oct 15;126:110681. doi: 10.1016/j.exger.2019.110681. Epub 2019 Aug 2. PMID 31382011
- [Background] Perez-Zepeda MU, Martinez-Velilla N, Kehler DS, Izquierdo M, Rockwood K, Theou O. The impact of an exercise intervention on frailty levels in hospitalised older adults: secondary analysis of a randomised controlled trial. Age Ageing. 2022 Feb 2;51(2):afac028. doi: 10.1093/ageing/afac028. PMID 35180287
- [Background] O'Brien MW, Kimmerly DS, Theou O. Impact of age and sex on the relationship between carotid intima-media thickness and frailty level in the Canadian Longitudinal Study of Aging. J Cardiol. 2023 Aug;82(2):140-145. doi: 10.1016/j.jjcc.2023.01.004. Epub 2023 Jan 20. PMID 36682711
- [Background] Church S, Rogers E, Rockwood K, Theou O. A scoping review of the Clinical Frailty Scale. BMC Geriatr. 2020 Oct 7;20(1):393. doi: 10.1186/s12877-020-01801-7. PMID 33028215
- [Background] O'Brien MW, Schwartz BD, Shivgulam ME, Daley WS, Frayne RJ, Kimmerly DS. Higher habitual lying time is inversely associated with vagal-related heart rate variability outcomes in younger adults. Appl Physiol Nutr Metab. 2023 Nov 1;48(11):876-881. doi: 10.1139/apnm-2023-0167. Epub 2023 Jul 10. PMID 37429038
- [Derived] Shivgulam ME, Dumont M, Ahmadi S, Courish M, Barrieau L, Cormier L, Theou O, Mekari S, O'Brien MW. Kinesiologist-delivered mobilization to mitigate inpatient frailty: A study protocol for a randomized controlled trial. Contemp Clin Trials. 2025 Dec 24;161:108204. doi: 10.1016/j.cct.2025.108204. Online ahead of print. PMID 41453522